CLINICAL TRIAL: NCT04257786
Title: Primary Cyto-reductive Surgery Vs Neo-adjuvant Chemotherapy (NAC) Followed by Surgery in Patients With Advanced Primary Epithelial Ovarian Cancer: A Pilot Randomized Study
Brief Title: Primary Cyto-reductive Surgery Vs Neo-adjuvant Chemotherapy (NAC) in Epithelial Ovarian Cancer
Acronym: ovarian cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ali hussien ali sayed, Specialist, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: epithelial ovarian cancer
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): 1ry surgery
  Interventions: Procedure: 1ry cyto-reductive surgery
- Group 2 (Active Comparator): Neoadjuvant Chemotherapy followed by surgery
  Interventions: Combination Product: Neoadjuvant chemotherapy followed by surgery

INTERVENTIONS:
Procedure: 1ry cyto-reductive surgery — 1ry surgery then chemotherapy
  Other Names: 1ry surgery
  Arms: Group 1
Combination Product: Neoadjuvant chemotherapy followed by surgery — chemotherapy then surgery
  Other Names: Neoadjuvant chemotherapy
  Arms: Group 2

SUMMARY:
Assessment of efficacy of primary cyto-reductive surgery in patients with advanced primary epithelial ovarian cancer in Comparison to patients receiving neo-adjuvant chemotherapy (NAC) followed by surgery in complete excision of the tumor reaching R0 without significant morbidity.

ELIGIBILITY:
Inclusion Criteria:

Female patients diagnosed with epithelial ovarian cancer (By histopathology)

Age ≥ 18 years old

Advanced defined as (stage 2D or more ) by surgical staging.

Performance status (PS) according to Eastern Cooperative Oncology Group (ECOG) ≤ 2

Chemotherapy naïve

Informed consent

Exclusion Criteria:

Patients previously received chemotherapy or radiotherapy to any part of the abdomen or pelvis.

Patients with uncontrolled infection.

Patients with active bleeding or conditions associated with high risk of bleeding.

contraindications for surgery

contraindications To chemotherapy - bevacizumab

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patient where complete resection of the tumor can be achieved | 3 month postoperative
  complete resection of the tumor

CONTACTS AND LOCATIONS:
Locations (1):
- Ali hussien Ali sayed, Asyut, Egypt

REFERENCES:
- [Derived] Abutaleb H, Hussien A, Khalaf M, Badary DM, Ismail AM, Hassanein S, AlGizawy S, Moustafa SAM, Farghaly RMM, Abdel-Kawi AF. Primary Cytoreductive Surgery Versus Neoadjuvant Chemotherapy Followed by Surgery in Patients with Advanced Primary Epithelial Ovarian Cancer in Low Resources Setting: A Randomized Clinical Trial. J Obstet Gynaecol India. 2025 Jun;75(3):199-205. doi: 10.1007/s13224-024-02061-w. Epub 2024 Nov 6. PMID 40584804